CLINICAL TRIAL: NCT05590052
Title: Bipolar Electrosurgery Versus Thermocautery in Circumcision With Safe Anesthetic Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DTH: 22003
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-09

CONDITIONS: Circumcision
Keywords: Circumcision; Electrosurgery; Thermocautery
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bipolar Electrosurgery group (n=60) (Active Comparator): Group A
  Interventions: Device: Bipolar Electrosurgery
- Thermocautery group (n=60) (Active Comparator): Group B
  Interventions: Device: Thermocautery

INTERVENTIONS:
Device: Bipolar Electrosurgery — Achievement of hemostasis using bipolar electrosurgery
  Arms: Bipolar Electrosurgery group (n=60)
Device: Thermocautery — achievement of hemostasis using thermocautery
  Arms: Thermocautery group (n=60)

SUMMARY:
Background: Circumcision is the most commonly performed surgical procedure done among the pediatric age group worldwide and is considered to be one of the oldest operations done. Circumcision should be performed properly with safe surgical techniques, with the least possibility of complications.

Objective: To compare bipolar electrosurgery versus thermocautery in the circumcision of infants under combined general and local anesthesia.

Patients and Methods: This prospective randomized comparative study was carried out on 110 infants who were candidates for elective circumcision under combined general and local anesthesia. Infants were randomly allocated into two equal groups (55 infants each); in group A, circumcised by bone-cutting forceps with cutting foreskin using a scalpel and achievement of hemostasis using bipolar electrosurgery, and in group B, circumcised by bone-cutting forceps with cutting foreskin and achievement of hemostasis using thermocautery.

ELIGIBILITY:
Inclusion Criteria:

* Infants of families who applied for circumcision
* Age from 1 to 12 months, of the male sex
* Infants should have normal preoperative laboratory investigations

Exclusion Criteria:

* Infants with congenital malformations especially hypospadias and epispadias, congenital inguinal hernia, and undescended testis
* Infants with acute penile infection, or excess suprapubic fat
* Infants with cardiovascular, neurological, respiratory, liver, renal, endocrine, blood, or immune diseases
* Allergy to any drug will be used in this study

Ages: 1 Month to 12 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Mean and Standard deviation of postoperative analgesic doses (mean±SD) | 72 hours after the end of the operation
  Number of analgesic doses given after the end of the operation

SECONDARY OUTCOMES:
Mean and Standard deviation of Operative duration (minutes) (mean±SD) | 2 minutes after the end of the operation
  Time from holding the penis till dresssing of the penis
Number of participants and Rate of Intraoperative complications | 2 minutes after the end of the operation
  Number of participants and Rate of: Tachycardia, Bradycardia, Laryngeal spasm, Hypoxia, Bleeding, Glans injury, and Vomiting.
Number of participants and Rate of Postoperative complications | 4 weeks after the end of the operation
  Number of participants and Rate of: Bleeding requiring surgical intervention, Penile edema, Wound infection, Meatal stenosis, and Trapped penis.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shaat, MD, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt